CLINICAL TRIAL: NCT04111510
Title: A Phase 2 Study of Autologous Tumor Infiltrating Lymphocytes (LN-145) in Patients With Pretreated Metastatic Triple Negative Breast Cancer
Brief Title: Autologous Tumor Infiltrating Lymphocytes in Patients With Pretreated Metastatic Triple Negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Iovance Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000025837
Record Dates: First submitted 2019-09-30; First posted 2019-10-01 (Actual); Results first posted 2024-02-23 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Metastatic Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Toll-Like Receptor 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LN-145 (Experimental): LN-145 will be delivered as a single therapy in patients with Metastatic Triple Negative Breast Cancer.
  Interventions: Drug: Tumor infiltrating lymphocytes (TIL) LN-145

INTERVENTIONS:
Drug: Tumor infiltrating lymphocytes (TIL) LN-145 — The TIL autologous therapy with LN-145 is comprised of the following steps:
  1. Tumor resection to provide the autologous tissue that serves as the source of the TIL cellular product;
  2. LN-145 investigational product production at a central Good Manufacturing Practice (GMP) facility;
  3. A 7-day nonmyeloablative lymphodepletion (NMA-LD) preconditioning regimen (hospitalization per institution standards);
  4. Infusion of the autologous LN-145 product on Day 0 (during inpatient hospitalization);
  5. Intravenous (IV) interleukin-2 (IL-2) administrations for up to six doses maximum (during inpatient hospitalization).

SUMMARY:
This study will investigate the safety and efficacy of TIL therapy in patients with metastatic TNBC who have progressed on at least one and no more than three prior systemic anticancer therapies.

DETAILED DESCRIPTION:
The primary aims of the study are:

* To evaluate the efficacy of autologous LN-145 as a single therapy in Metastatic Triple Negative Breast Cancer (TNBC) patients by determining the objective response rate (ORR), using the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, as assessed by the Investigator.
* To characterize the safety profile of tumor infiltrating lymphocytes (TIL) as a single therapy in Metastatic Triple Negative Breast Cancer patients as measured by the incidence of Grade ≥ 3 treatment-emergent adverse events (TEAEs).

The secondary aims of the study are:

• To further evaluate the efficacy of autologous LN-145 as a single therapy in Metastatic Triple Negative Breast Cancer patients using complete response duration of response (DOR), disease control rate (DCR), and progression-free survival (PFS), using RECIST 1.1, as assessed by the Investigator, overall survival (OS) and (CR) rate.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand the requirements of the study. Specifically, the patient has to provide written informed consent (as evidenced by signature on an ICF approved by the Yale Human Investigation Committee (HIC).
* All patients must have a triple negative metastatic breast cancer (Estrogen Receptor negative, Progesterone Receptor negative, HER2 negative) as defined by the 2018 ASCO CAP guidelines.
* Patients must have a confirmed diagnosis of metastatic triple negative breast cancer (Stage IV) histologically confirmed as per American Joint Committee on Cancer [AJCC] staging system).
* Patients must have had at least one and no more than three prior lines of systemic anticancer therapies for metastatic disease.
* Patients must have disease progression from the last line of therapy.
* Patients must have at least one resectable lesion of a minimum 1.5 cm in diameter (or aggregate of 1.5 cm if multiple lesions are sampled) post-resection for TIL investigational product production.
* Patients must have remaining measurable disease as defined by RECIST 1.1 following tumor resection for TIL manufacturing
* Patients must be ≥ 18 years of age at the time of consent.
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1, and an estimated life expectancy of ≥ 3 months in the opinion of the Investigator.
* Female patients of childbearing potential or female partners of childbearing potential of male participants, must be willing to practice an approved method of birth control during treatment and for 12 months after receiving all protocol-related therapy.
* Patients must have the following hematologic parameters:

  * Absolute neutrophil count (ANC) ≥ 1000/mm3;
  * Hemoglobin ≥ 9.0 g/dL;
  * Platelet count ≥ 100,000/mm3
* Patients must have adequate organ function.
* Patients must be seronegative for the human immunodeficiency virus (HIV1 and HIV2).
* Patients must have a washout period of 21 days from last anticancer therapy prior to the first study treatment (ie, start of NMA LD).
* Palliative radiation therapy: prior external beam radiation is allowed provided all radiation-related toxicities are resolved to Grade 1 or baseline;

  * The tumor lesion(s) being assessed as target for response via RECIST 1.1 must be outside of the radiation portal (however, if within the portal, they must have demonstrated progression);
  * Surgery/pre-planned procedure: previous surgical procedure(s) is permitted provided that wound healing has occurred, all complications have resolved, and at least 14 days have elapsed (for major operative procedures) prior to the tumor resection.
* Patients must have recovered from all prior anticancer treatment-related adverse events (TRAEs) to Grade ≤ 1 (per Common Terminology Criteria for Adverse Events [CTCAE], version 5.0).
* Patients must have provided written authorization for use and disclosure of protected health information.
* Must be able and willing to comply with the study visit schedule and protocol requirements including long-term follow-up (LTFU).

Exclusion Criteria:

* Patients who have received an organ allograft or prior cell transfer therapy within the past 20 years that included a nonmyeloablative or myeloablative chemotherapy regimen.
* Patients with symptomatic and/or untreated brain metastases:
* Patients who are on systemic steroid therapy except for those requiring steroid for management of adrenal insufficiency.
* Patients who are pregnant or breastfeeding.
* Patients who have active medical illness(es) that would pose increased risk for study participation
* Patients who have received a live or attenuated vaccination within 28 days prior to the start of NMA-LD.
* Patients who have any form of primary immunodeficiency (such as severe combined immunodeficiency disease [SCID] and acquired immune deficiency syndrome [AIDS]).
* Patients with a history of hypersensitivity to any component of the study drugs.
* Patients who have a left ventricular ejection fraction (LVEF) < 45% or who are New York Heart Association (NYHA) Class II or higher.
* Patients who have obstructive or restrictive pulmonary disease and have a documented FEV1 (forced expiratory volume in 1 second) ≤ 60% of predicted normal.
* Patients who have had another primary malignancy within the previous 3 years (except for curatively treated localized malignancy that has not required treatment for greater than 1 year.
* Participation in another clinical study with an investigational product within 21 days of the initiation of NMA-LD treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-12-23 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hurwitz, MD, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Gautam N, Elleson KM, Ramamoorthi G, Czerniecki BJ. Current State of Cell Therapies for Breast Cancer. Cancer J. 2022 Jul-Aug 01;28(4):301-309. doi: 10.1097/PPO.0000000000000607. PMID 35880940

RESULTS

PARTICIPANT FLOW:
Groups:
- LN-145: LN-145 will be delivered as a single therapy in patients with Metastatic Triple Negative Breast Cancer.
  Tumor infiltrating lymphocytes (TIL) LN-145: The TIL autologous therapy with LN-145 is comprised of the following steps:
  1. Tumor resection to provide the autologous tissue that serves as the source of the TIL cellular product;
  2. LN-145 investigational product production at a central Good Manufacturing Practice (GMP) facility;
  3. A 7-day nonmyeloablative lymphodepletion (NMA-LD) preconditioning regimen (hospitalization per institution standards);
  4. Infusion of the autologous LN-145 product on Day 0 (during inpatient hospitalization);
  5. Intravenous (IV) interleukin-2 (IL-2) administrations for up to six doses maximum (during inpatient hospitalization).
Period: Overall Study
Arm/Group | LN-145
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | LN-145
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: To evaluate the efficacy of autologous LN-145 as a single therapy in Metastatic Triple Negative Breast Cancer (TNBC) patients by determining the objective response rate (ORR), using the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, as assessed by the Investigator. Upon results entry, the time frame was updated to reflect the latest time point that a participant was assessed for ORR in the study.
Time Frame: Up to 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | LN-145
Number analyzed (Participants) | 6
Participants
  complete response (CR) | 0
  partial response (PR) | 1
  stable disease (SD) | 1
  progressive disease (PD) | 4

2. Primary Outcome: Safety Profile
Description: To characterize the safety profile of tumor infiltrating lymphocytes (TIL) as a single therapy in Metastatic Triple Negative Breast Cancer patients as measured by the incidence of Grade ≥ 3 treatment-emergent adverse events (TEAEs). Incidence is presented as a count of participants that experienced at least 1 TEAE of Grade ≥ 3.
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | LN-145
Number analyzed (Participants) | 6
Participants | 3

3. Secondary Outcome: Duration of Response (DOR) in Days
Description: To evaluate the efficacy of autologous LN-145 as a single therapy in Metastatic Triple Negative Breast Cancer patients in participants that have a clinical response (either partial response (PR) or complete response (CR)) using duration of response (DOR), using RECIST 1.1, as assessed by the Investigator will be used.
Time Frame: Up to 3 years
Population: Only assessed in participants that had a PR. Only one participant had a PR. Method of dispersion was not collected as was only one participant.
Measure: Number; unit: days
Arm/Group | LN-145
Number analyzed (Participants) | 1
days | 79

4. Secondary Outcome: Disease Control Rate (DCR)
Description: To evaluate the efficacy of autologous LN-145 as a single therapy in Metastatic Triple Negative Breast Cancer patients using disease control rate (DCR), using RECIST 1.1, as assessed by the Investigator will be used. Percentage of patients whose disease shrinks or remains stable over a certain time period.
Time Frame: Up to 3 years
Measure: Number; unit: percentage of participants
Arm/Group | LN-145
Number analyzed (Participants) | 6
percentage of participants | 66.6

5. Secondary Outcome: Progression-free Survival (PFS)
Description: To evaluate the efficacy of autologous LN-145 as a single therapy in Metastatic Triple Negative Breast Cancer patients, median progression-free survival (PFS) days, using RECIST 1.1, as assessed by the Investigator will be used.
Time Frame: Up to 3 years
Measure: Median (Standard Deviation); unit: days
Arm/Group | LN-145
Number analyzed (Participants) | 6
days | 46.5 (19.8)

6. Secondary Outcome: Overall Survival (OS)
Description: To evaluate the efficacy of autologous LN-145 as a single therapy in Metastatic Triple Negative Breast patients overall survival (OS) median days will be used.
Time Frame: Up to 3 years
Measure: Median (Standard Deviation); unit: days
Arm/Group | LN-145
Number analyzed (Participants) | 6
days | 156.5 (66.8)

7. Secondary Outcome: Complete Response (CR)
Description: To evaluate the efficacy of autologous LN-145 as a single therapy in Metastatic Triple Negative Breast patients complete response, using RECIST 1.1, as assessed by the Investigator will be used. The number of participants with a complete response.
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | LN-145
Number analyzed (Participants) | 6
Participants | 0

ADVERSE EVENTS:
Time Frame: Up to 3 years
Arm/Group | LN-145
All-Cause Mortality (participants affected / at risk) | 6/6
Serious Adverse Events (participants affected / at risk) | 4/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LN-145 (N=6)
Neutrophil count decreased (Investigations) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Fatigue (General disorders) | 1 (2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LN-145 (N=6)
Anemia (Blood and lymphatic system disorders) | 4 (8)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (4)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 4 (5)
White blood cell count decreased (Blood and lymphatic system disorders) | 4 (10)
Lymphopenia (Blood and lymphatic system disorders) | 4 (15)
Platelet count decreased (Blood and lymphatic system disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 5 (5)
Nausea (Gastrointestinal disorders) | 5 (7)
Diarrhea (Gastrointestinal disorders) | 4 (7)
Loss of appetite (Gastrointestinal disorders) | 1 (1)
Intermittent Emesis (Gastrointestinal disorders) | 2 (2)
Fever (General disorders) | 5 (7)
Chills (General disorders) | 2 (2)
Fatigue (General disorders) | 3 (4)
Rigors (General disorders) | 4 (5)
Pain (General disorders) | 2 (5)
Weight Gain (General disorders) | 1 (1)
Infection (General disorders) | 2 (2)
Dehydration (General disorders) | 1 (1)
Hair loss (General disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 2 (2)
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 3 (4)
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 1 (1)
Blood bilirubin increased (Metabolism and nutrition disorders) | 2 (2)
CPK increased (Metabolism and nutrition disorders) | 1 (2)
Creatinine increased (Metabolism and nutrition disorders) | 1 (1)
Lipase increased (Metabolism and nutrition disorders) | 1 (1)
Serum amylase increased (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (6)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (3)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Headache (Nervous system disorders) | 4 (6)
Confusion (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Hand tremor (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
General edema (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Thrombocytopenia (Vascular disorders) | 4 (11)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-10): https://cdn.clinicaltrials.gov/large-docs/10/NCT04111510/Prot_SAP_000.pdf